CLINICAL TRIAL: NCT04409769
Title: Evaluation of the Tolerance of Anti-MRSA Betalactamines (Ceftaroline / Ceftobiprole) in the Management of BJI / PJI: a Retrospective Study in a Reference Center
Brief Title: Evaluation of the Tolerance of Ceftaroline and Ceftobiprole in the Management of BJI / PJI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20-157
Record Dates: First submitted 2020-05-12; First posted 2020-06-01 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Bone and Joint Infection; Antibiotic Reaction
Keywords: bone and joint infection; prosthesis joint infection; adverse event; ceftaroline; ceftobiprole
MeSH Terms: interventions — ceftobiprole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Description of use of ceftaroline and ceftobiprole: description of patients and their PJI/BJI,conditions of use, adverse event
  Interventions: Other: Description of use of ceftaroline and ceftobiprole

INTERVENTIONS:
Other: Description of use of ceftaroline and ceftobiprole — Ceftaroline and ceftobiprole are the only betalactam active on methicillin-resistant staphylococci. Description of condition of use of thoses antibiotics in PJI and BJI

SUMMARY:
Staphyloccous aureus and coagulase negative staphylocci are responsible of a large marjority of PJI. Regarding the high rate of methicillin resistance, current guidelines recommend the use of a glycopeptide, and most frequently vancomycin, as the anti-gram positive agent in empirical therapy, while awaiting the microbiological results. Vancomycin is not considered as a safe antibiotic, and daptomycin is frequently an alternative option.

Ceftaroline and ceftobiprole are the only betalactam active on methicillin-resistant staphylococci. As some data report a synergistic activity with daptomycin, they could be an option in pandrug-resistant staphylococci BJI, but their use if off label in this indication.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a PJI or BJI treated whith ceftaroline and/or ceftobiprole

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had a PJI or BJI treated whith ceftaroline and/or ceftobiprole treated at CRIOAc Lyon
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of use of ceftaroline and ceftobiprole : patients | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  type of patients: age, CMI
Evaluation of use of ceftaroline: dosage | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  dosage,duration
Evaluation of use of ceftaroline : PJI/BJI | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  description of the PJI/BJI treated by ceftaroline : presence of knee or hip prosthesis, evolution between prosthesis placement and the onset of symptoms, gateway to infection
Evaluation of use of ceftobiprole: dosage | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  dosage, duration
Evaluation of use of ceftobiprole: PJI/BJI | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  description of the PJI/BJI treated by ceftobiprole : presence of knee or hip prosthesis, evolution between prosthesis placement and the onset of symptoms, gateway to infection
rate of failure under ceftaroline | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin
rate of failure under ceftobiprole | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

SECONDARY OUTCOMES:
Treatment-related adverse events | 2 months
  description of adverse event under ceftaroline and/or ceftobiprole as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr